CLINICAL TRIAL: NCT03362034
Title: Chairside Time and Accuracy of Indirect Bonding of Orthodontic Attachments Using Double Versus Single Transfer Tray: A Randomized Controlled Trial
Brief Title: Chairside Time and Accuracy of Indirect Bonding of Orthodontic Attachments Using Double Versus Single Transfer Tray
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohamed essam, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CEBC-CU-2017-11-14
Record Dates: First submitted 2017-11-21; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Orthodontic Appliance Complication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single transfer tray (Active Comparator)
  Interventions: Device: single transfer tray
- double transfer trays (Experimental)
  Interventions: Device: double transfer trays

INTERVENTIONS:
Device: double transfer trays — double trays one soft and one hard
  Arms: double transfer trays
Device: single transfer tray — single soft tray
  Arms: single transfer tray

SUMMARY:
compare the chairside time and the accuracy of transferring attachments between single and double sheets vacuum tray techniques during indirect bonding of orthodontic attachments using superimposition on computer software

ELIGIBILITY:
Inclusion Criteria:

1. Patient with maxillary full set of teeth and undergoing fixed orthodontic treatment.
2. Good oral hygiene.
3. Mild to moderate crowding.

Exclusion Criteria:

1. Patients with partially erupted teeth in the maxillary arch.
2. Signs of caries, large restorations or abnormalities of crown morphology.
3. The need of banding.
4. Bad oral hygiene measures.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Chairside time of brackets bonding | an average of 30 minutes
  using Stop watch

SECONDARY OUTCOMES:
Accuracy of orthodontic attachments transfer | one day after bonding
  linear (mm) scale using geomagic software
Accuracy of orthodontic attachments transfer | one day after bonding
  angular (degrees) scale using geomagic software

OTHER OUTCOMES:
immediate Bond failure | immediately after bonding
  number of debonded attachments using hand instrument pressure